CLINICAL TRIAL: NCT03835676
Title: Effects of Treprostinil on Right Ventricular Structure and Function in Patients With Pulmonary Arterial Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Magdi H. Yacoub (Other)
Responsible Party: Sponsor-Investigator, Magdi H. Yacoub, Principal Investigator - Sir. Prof., OM FRS, Magdi Yacoub Heart Foundation
Organization: Magdi Yacoub Heart Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Treprostinil RV
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; Right ventricular function
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Intervention Model Description: In a group of patients with PAH treated with treprostinil, the current study aims to investigate the effect of treatment on RV structure and function; and correlate changes in RV structure and function with: WHO class, Six-minute walk test, Quality of life (QoL), and Pre-specified biomarkers (NT-ProBNP, Tissue growth factor-B BNP, and Profibrotic markers)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary hypertension treated with Treprostinil (Experimental): Thirty patients who will be treated with Treprostinil.
  Interventions: Drug: Treprostinil

INTERVENTIONS:
Drug: Treprostinil — After inclusion and baseline measurements, patients will receive treprostinil in addition to background therapy for 24 months. Follow-up assessment will include:
  * Clinical, echocardiographic, laboratory assessments will be repeated at 1, 3, 6, 12, 18, and 24 month (or when there is clinical indication)
  * CMR will be performed at 6 monthly intervals for 2 years.
  * Peak power output at 6,12, 18 and 24 month
  * Right-side cardiac catheterization will be performed at 6, 12 , 18 and 24 months (or when there is clinical indication)
  Other Names: Remodulin

SUMMARY:
In a group of patients with PAH treated with treprostinil, the current study aims to investigate the effect of treatment on RV structure and function; and correlate changes in RV structure and function with: World Health Organisation (WHO) class, Six-minute walk test, Quality of life (QoL), and Pre-specified biomarkers (N-terminal B-type natriuretic peptide (NT-ProBNP), Tissue growth factor-B B-type natriuretic peptide BNP, and Profibrotic markers)

DETAILED DESCRIPTION:
A) Right ventricle (RV) in pulmonary hypertension

RV failure is the main cause of death in patients with pulmonary arterial hypertension (PAH), and the ability of the RV to adapt to the progressive increase in pulmonary vascular resistance associated with changes to the pulmonary vasculature in PAH is the main determinant of a patient's functional capacity and survival.

The response of the right ventricle (RV) to the increase in afterload produced by the pulmonary vascular changes characteristic of PAH is the key factor in the development of symptoms and in determining survival. Structurally, rising systolic and diastolic ventricular pressures increase diastolic and systolic stretch on the RV wall, which leads initially to an increase in muscle mass (adaptive hypertrophy) due to increased protein synthesis and an increase in cardiomyocyte size through the addition of sarcomeres. However, the RV cannot maintain adaptive hypertrophy in the face of sustained pressure overload, and eventually there is a transition to dilatation. At this stage there is no further increase, or even a decrease, in RV contractility, despite a further increase in load. One consequence of RV dilatation is an increase in wall tension, which increases myocardial oxygen demand and simultaneously decreases RV perfusion, leading to further compromised contractility and dilatation.

The exact mechanisms leading to the development of RV failure in patients with PAH are still unclear. Several mechanisms have been hypothesized: RV myocardial ischaemia, microvascular endothelial cell dysfunction, and myocyte apoptosis. In severe end-stage PAH, the RV changes its shape from the normal conformation to a more spherical one, and RV wall stress increases because RV wall thickness does not increase proportionally.

Given the importance of the RV in PAH, preservation and improvement of its function should be important aspects of therapy; however, there are currently few data specifically related to this aspect of treatment response.

B) Vasodilator therapy and RV in pulmonary hypertension Although RV failure is the main cause of death in patients with pulmonary arterial hypertension (PAH), there is insufficient data about the effects of PAH treatment on RV geometry and function mainly because the RV assessment has been hampered by its complex crescentic shape, large infundibulum, and its trabecular nature. . This is specifically true for vasodilator therapies. Such therapies may affect the RV via direct cardiac-specific effects or indirect effects by reducing RV load. In a meta-analysis of clinical studies of PAH-specific therapies, active treatment was associated with a reduction in pulmonary vascular resistance which was accompanied by a decrease in pulmonary artery pressure, and an increase in stroke volume, but without an increase in contractility, suggesting that current PAH therapies have predominantly pulmonary vasodilating effects and have limited cardiac-specific effects. In a study of epoprostenol therapy, beneficial effects on RV structure and function (RV dilatation, curvature of the interventricular septum and maximal tricuspid regurgitant jet velocity) compared with placebo were reported following 12 weeks of treatment, with change in 6-min walk distance between baseline and 12 weeks being inversely related to the change in diastolic eccentricity index and pericardial effusion size. Such improvements may contribute to the clinical improvement and prolonged survival observed with epoprostenol in other studies.

Other evidence of improvements in RV parameters has come from descriptive studies using a number of PAH-specific therapies; however, these generally include a small number of patients, and this, together with the fact that such studies evaluated different parameters (both in terms of functional parameters and measures of RV size/mass), makes the assessment of results difficult. longer term studies of epoprostenol have not shown a positive treatment effect on RV size/mass although without a comparator arm it is not possible to determine whether long-term therapy slowed down the rate of RV hypertrophy or dilatation.

Overall, therefore, the effects of PAH-specific therapies on RV function remain to be fully investigated.

C) Treprostinil Treprostinil is a tricyclic benzindene analogue of prostacyclin, and has as such similar anti-platelet and vasodilatory actions, including acute pulmonary vasodilation.

Treprostinil, a stable prostacyclin analog, has similar pharmacologic effects to epoprostenol, However, in contrast to epoprostenol, treprostinil is chemically stable at room temperature and neutral 'power of hydrogen' (pH) and has a longer half-life (elimination half-life of 4.5 h with distribution half-life of 40 min, compared with 2 to 3 min for epoprostenol) permitting continuous subcutaneous infusion (16). Treprostinil has been shown in a large multicenter randomized controlled trial to improve exercise capacity, clinical state, functional class, pulmonary hemodynamics, and quality of life in patients with pulmonary arterial hypertension.

D) Assessment of RV with cardiac magnetic resonance imaging Currently, the most widely used noninvasive techniques are echocardiography and cardiac magnetic resonance imaging), and a number of potential indicators assessed using these methods have been proposed. Cardiac magnetic resonance imaging provides a higher spatial resolution, and is not limited by factors affecting echocardiography (e.g. acoustic window). Cardiac magnetic resonance imaging allows for the visualisation and measurement of complex three-dimensional geometry and it is therefore particularly suited to the complex morphology of the RV. Precise, noninvasive assessment of cardiac volumes and function is possible, without the need for geometric approximations, while assessments such as flow measurements in the heart and great vessels using techniques such as cine phase-contrast provide more comprehensive data on cardiac function than echocardiography.

ELIGIBILITY:
* Inclusion Criteria:

  * PAH defined as a mean pulmonary artery pressure >25 mmHg on right heart catheterization at rest in the setting of a normal pulmonary arterial wedge pressure ≤15 mm Hg
  * PAH that is idiopathic, familial, or associated with connective tissue disease.
  * WHO class III or class IV despite the use of Endothelin receptor antagonists (ERA) and/or phosphodiesterase-5 inhibitors
  * Age > 18 years
  * Sinus rhythm
* Exclusion Criteria:

  * Patients with PAH associated with HIV infection, portal hypertension, congenital heart disease, schistosomiasis, chronic haemolytic anaemia
  * Patients with pulmonary hypertension due to veno-occlusive disease and/or pulmonarycapillary haemangiomatosis, thromboembolism.
  * Patients with left side heart disease that may contribute to pulmonary hypertension. Those patients are identified by having pulmonary wedge pressure >15 mmHg or elevated Left Ventricle (LV) end-diastolic pressure
  * Patients who are severely disabled and will not be able to complete the study
  * Patients with significant lung disease as shown by forced vital capacity (FVC) < 70% predicted, or forced expiratory volume at one second (FEV1)/FVC < 50% - Life expectancy <1 year due to severe PAH or any other forms of terminal disease.
  * Pregnant women
  * Refusal to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Treprostinil effects on right ventricular structure and function using echocardiography | through study completion, an average of 5 years
  Assessment of RV structure and function by echocardiography
Assessment of Treprostinil effects on right ventricular structure and function using Cardiac Magnetic Resonance Imaging (CMR). | through study completion, an average of 5 years
  Assessment of RV structure and function by cardiac magnetic resonance imaging (CMR).

SECONDARY OUTCOMES:
Correlate changes in RV structure and function with World Health Organisation (WHO) Class. | through study completion, an average of 5 years
  correlate changes in RV structure and function with the WHO class.
Correlate changes in RV structure and function with the Six-minute walk test results | through study completion, an average of 5 years
  correlate changes in RV structure and function with the Six-minute walk test results
Correlate changes in RV structure and function with QoL | through study completion, an average of 5 years
  correlate changes in RV structure and function with the Quality of life (QoL)
Correlate changes in RV structure and function with prespecified biomarkers | through study completion, an average of 5 years
  correlate changes in RV structure and function with the Pre-specified biomarkers (NT-ProBNP, Tissue growth factor-B BNP, and Profibrotic markers)

CONTACTS AND LOCATIONS:
Overall Officials: Magdi H Yacoub, OM FRS, Study Chair — Magdi Yacoub Heart Foundation - Aswan Heart Centre
Locations (1):
- Aswan Heart Centre - Magdi Yacoub Heart Foundation, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Handoko ML, de Man FS, Allaart CP, Paulus WJ, Westerhof N, Vonk-Noordegraaf A. Perspectives on novel therapeutic strategies for right heart failure in pulmonary arterial hypertension: lessons from the left heart. Eur Respir Rev. 2010 Mar;19(115):72-82. doi: 10.1183/09059180.00007109. PMID 20956170
- [Background] Benza R, Biederman R, Murali S, Gupta H. Role of cardiac magnetic resonance imaging in the management of patients with pulmonary arterial hypertension. J Am Coll Cardiol. 2008 Nov 18;52(21):1683-92. doi: 10.1016/j.jacc.2008.08.033. PMID 19007687
- [Background] Boxt LM, Katz J, Kolb T, Czegledy FP, Barst RJ. Direct quantitation of right and left ventricular volumes with nuclear magnetic resonance imaging in patients with primary pulmonary hypertension. J Am Coll Cardiol. 1992 Jun;19(7):1508-15. doi: 10.1016/0735-1097(92)90611-p. PMID 1593046
- [Background] Quaife RA, Chen MY, Lynch D, Badesch DB, Groves BM, Wolfel E, Robertson AD, Bristow MR, Voelkel NF. Importance of right ventricular end-systolic regional wall stress in idiopathic pulmonary arterial hypertension: a new method for estimation of right ventricular wall stress. Eur J Med Res. 2006 May 5;11(5):214-20. PMID 16723296
- [Background] McLaughlin VV, Archer SL, Badesch DB, Barst RJ, Farber HW, Lindner JR, Mathier MA, McGoon MD, Park MH, Rosenson RS, Rubin LJ, Tapson VF, Varga J; American College of Cardiology Foundation Task Force on Expert Consensus Documents; American Heart Association; American College of Chest Physicians; American Thoracic Society, Inc; Pulmonary Hypertension Association. ACCF/AHA 2009 expert consensus document on pulmonary hypertension a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents and the American Heart Association developed in collaboration with the American College of Chest Physicians; American Thoracic Society, Inc.; and the Pulmonary Hypertension Association. J Am Coll Cardiol. 2009 Apr 28;53(17):1573-619. doi: 10.1016/j.jacc.2009.01.004. No abstract available. PMID 19389575
- [Background] Hinderliter AL, Willis PW 4th, Long W, Clarke WR, Ralph D, Caldwell EJ, Williams W, Ettinger NA, Hill NS, Summer WR, de Biosblanc B, Koch G, Li S, Clayton LM, Jobsis MM, Crow JW. Frequency and prognostic significance of pericardial effusion in primary pulmonary hypertension. PPH Study Group. Primary pulmonary hypertension. Am J Cardiol. 1999 Aug 15;84(4):481-4, A10. doi: 10.1016/s0002-9149(99)00342-2. PMID 10468096
- [Background] Barst RJ, Rubin LJ, McGoon MD, Caldwell EJ, Long WA, Levy PS. Survival in primary pulmonary hypertension with long-term continuous intravenous prostacyclin. Ann Intern Med. 1994 Sep 15;121(6):409-15. doi: 10.7326/0003-4819-121-6-199409150-00003. PMID 8053614
- [Background] Barst RJ, Rubin LJ, Long WA, McGoon MD, Rich S, Badesch DB, Groves BM, Tapson VF, Bourge RC, Brundage BH, Koerner SK, Langleben D, Keller CA, Murali S, Uretsky BF, Clayton LM, Jobsis MM, Blackburn SD, Shortino D, Crow JW; Primary Pulmonary Hypertension Study Group. A comparison of continuous intravenous epoprostenol (prostacyclin) with conventional therapy for primary pulmonary hypertension. N Engl J Med. 1996 Feb 1;334(5):296-301. doi: 10.1056/NEJM199602013340504. PMID 8532025
- [Background] Sebbag I, Rudski LG, Therrien J, Hirsch A, Langleben D. Effect of chronic infusion of epoprostenol on echocardiographic right ventricular myocardial performance index and its relation to clinical outcome in patients with primary pulmonary hypertension. Am J Cardiol. 2001 Nov 1;88(9):1060-3. doi: 10.1016/s0002-9149(01)01995-6. No abstract available. PMID 11704014
- [Background] Roeleveld RJ, Vonk-Noordegraaf A, Marcus JT, Bronzwaer JG, Marques KM, Postmus PE, Boonstra A. Effects of epoprostenol on right ventricular hypertrophy and dilatation in pulmonary hypertension. Chest. 2004 Feb;125(2):572-9. doi: 10.1378/chest.125.2.572. PMID 14769740
- [Background] Bristow MR, Zisman LS, Lowes BD, Abraham WT, Badesch DB, Groves BM, Voelkel NF, Lynch DM, Quaife RA. The pressure-overloaded right ventricle in pulmonary hypertension. Chest. 1998 Jul;114(1 Suppl):101S-106S. doi: 10.1378/chest.114.1_supplement.101s. No abstract available. PMID 9676654
- [Background] Vachiery JL, Hill N, Zwicke D, Barst R, Blackburn S, Naeije R. Transitioning from i.v. epoprostenol to subcutaneous treprostinil in pulmonary arterial hypertension. Chest. 2002 May;121(5):1561-5. doi: 10.1378/chest.121.5.1561. PMID 12006444
- [Background] McNulty MJ, Sailstad JM, Steffen RP. The pharmacokinetics and pharmacodynamics of the prostacyclin analog 15AU81 in the anesthetized beagle dog. Prostaglandins Leukot Essent Fatty Acids. 1993 Feb;48(2):159-66. doi: 10.1016/0952-3278(93)90105-6. PMID 8446654
- [Background] Laliberte K, Arneson C, Jeffs R, Hunt T, Wade M. Pharmacokinetics and steady-state bioequivalence of treprostinil sodium (Remodulin) administered by the intravenous and subcutaneous route to normal volunteers. J Cardiovasc Pharmacol. 2004 Aug;44(2):209-14. doi: 10.1097/00005344-200408000-00010. PMID 15243302
- [Background] Simonneau G, Barst RJ, Galie N, Naeije R, Rich S, Bourge RC, Keogh A, Oudiz R, Frost A, Blackburn SD, Crow JW, Rubin LJ; Treprostinil Study Group. Continuous subcutaneous infusion of treprostinil, a prostacyclin analogue, in patients with pulmonary arterial hypertension: a double-blind, randomized, placebo-controlled trial. Am J Respir Crit Care Med. 2002 Mar 15;165(6):800-4. doi: 10.1164/ajrccm.165.6.2106079. PMID 11897647
- [Background] Gomberg-Maitland M, Tapson VF, Benza RL, McLaughlin VV, Krichman A, Widlitz AC, Barst RJ. Transition from intravenous epoprostenol to intravenous treprostinil in pulmonary hypertension. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1586-9. doi: 10.1164/rccm.200505-766OC. Epub 2005 Sep 8. PMID 16151039
- [Background] Kovacs G, Reiter G, Reiter U, Rienmuller R, Peacock A, Olschewski H. The emerging role of magnetic resonance imaging in the diagnosis and management of pulmonary hypertension. Respiration. 2008;76(4):458-70. doi: 10.1159/000158548. Epub 2008 Nov 12. PMID 19018164
- [Background] Towbin JA. Scarring in the heart--a reversible phenomenon? N Engl J Med. 2007 Oct 25;357(17):1767-8. doi: 10.1056/NEJMcibr075397. No abstract available. PMID 17960018
- [Background] Zannad F, Alla F, Dousset B, Perez A, Pitt B. Limitation of excessive extracellular matrix turnover may contribute to survival benefit of spironolactone therapy in patients with congestive heart failure: insights from the randomized aldactone evaluation study (RALES). Rales Investigators. Circulation. 2000 Nov 28;102(22):2700-6. doi: 10.1161/01.cir.102.22.2700. PMID 11094035
- [Background] Morais P, Marchi A, Bogaert JA, Dresselaers T, Heyde B, D'hooge J, Bogaert J. Cardiovascular magnetic resonance myocardial feature tracking using a non-rigid, elastic image registration algorithm: assessment of variability in a real-life clinical setting. J Cardiovasc Magn Reson. 2017 Feb 17;19(1):24. doi: 10.1186/s12968-017-0333-y. PMID 28209163